CLINICAL TRIAL: NCT00250224
Title: Prostate Localization During Radiotherapy Using a Ni-Ti Stent and Electronic Portal Imaging - Protocol II
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: stent02
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2005-09

CONDITIONS: Prostatic Neoplasms
Keywords: Radiotherapy; image guided; marker
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stent (Experimental)
  Interventions: Device: Radiotherapy stent

INTERVENTIONS:
Device: Radiotherapy stent

SUMMARY:
A new method for localization of the prostate during external beam radiotherapy. The method is based on insertion of a new thermo-expandable Ni-Ti stent. The radiological properties of the stent are used for precise prostate localization during treatment using electronic portal images

DETAILED DESCRIPTION:
Inclusion criteria's in the study were 1) Patients should present with histological verified local or locally advanced PC (stage T2b to T3b, N0, M0; UICC 1992 classification was used). 2) Patients should consequently be candidates for intended curative radiotherapy. Prostatic work up is done before inclusion in the study. A new prostatic Nickel - Titanium stent is placed in the prostatic urethra one week prior to the radiotherapy planning CT using a flexible cystoscope to insert the stent under urethral anaesthesia. The stent is then flushed with hot water (60 degrees Celsius). The hot water expands the stent collar, thereby locking the stent in place. Correct positioning of the stent is secured visually on retraction of the scope. Radiotherapy of prostate is given to a mean dose of 70 (department standard regime). Treatment are given with daily fractions of 2 Gy using a combination of 6 MV and 18 MV X-ray fields using isocentric 3D conformal treatment plan, consisting of three MLC conformal radiation fields (One anterior and two lateral wedged fields). This was assumed to be the optimal treatment plan. A pair of orthogonal 15 cm x 15 cm isocenter setup fields was added to the plan. The orthogonal fields are used to obtain pairs of electronic portal images. Electronic portal images are recorded using a Varian As500 electronic portal imaging device (EPID). The images are used to determine the 3D reference position of the stent. The image pairs of the stent were taken at eight treatment sessions in each patient (Session number 1,2,3,6,11,21,22 and 23). From each orthogonal set of images the 3D position of both the stent and the symphysis (pubic bone) are determined. Positions are calculated using orthogonal reconstruction. A control CT scan is made before treatment session number 21 to verify the intra prostatic position of the stent. The intra prostatic position of the stent is also verified during removal of the stent three months after radiation therapy. Before removal the stent was flushed with water at 10 degrees Celsius. When cooled with 10°C cold water, the stent became super soft, and can easily be removed as a twisted wire.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should present with histological verified local or locally advanced PC (stage T2b to T3b, N0, M0; UICC 1992 classification was used).
2. Patients should consequently be candidates for intended curative radiotherapy -

Exclusion Criteria:

dislocation or removal of stent

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-01; Primary Completion 2009-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
stent in situ during radiotherapy | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Carl, PhD, Study Chair — Dept medical Physics, Oncology
Locations (1):
- Dept of oncology, Aalborg, North Denmark, Denmark

REFERENCES:
- [Background] Carl J, Sander L. Five-year follow-up using a prostate stent as fiducial in image-guided radiotherapy of prostate cancer. Acta Oncol. 2015 Jun;54(6):862-7. doi: 10.3109/0284186X.2014.987355. Epub 2014 Dec 24. PMID 25539443
- [Background] Sander L, Langkilde NC, Holmberg M, Carl J. MRI target delineation may reduce long-term toxicity after prostate radiotherapy. Acta Oncol. 2014 Jun;53(6):809-14. doi: 10.3109/0284186X.2013.865077. Epub 2013 Dec 20. PMID 24358954
- [Background] Carl J, Nielsen J, Holmberg M, Larsen EH, Fabrin K, Fisker RV. Clinical results from first use of prostate stent as fiducial for radiotherapy of prostate cancer. Acta Oncol. 2011 May;50(4):547-54. doi: 10.3109/0284186X.2010.541935. Epub 2010 Dec 21. PMID 21174520